CLINICAL TRIAL: NCT04366635
Title: Evaluation of the Effectiveness of the Mineralized Plasmatic Matrix and Tricalcium Phosphate Graft Application After Mandibular Impacted Third Molar Surgery in Terms of Periodontal and Osseous Healing Distal to the Second Molar
Brief Title: Evaluation of Two Different Grafting Techniques After Mandibular Impacted Third Molar Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Konya Necmettin Erbakan Üniversitesi (Other)
Responsible Party: Principal Investigator, Ali Kılınç, Research Assistant, Konya Necmettin Erbakan Üniversitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KonyaNEU1
Record Dates: First submitted 2020-04-26; First posted 2020-04-29 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Periodontal Pocket; Impacted Third Molar Tooth; Impacted Teeth With Abnormal Position
Keywords: Mineralized Plasmatic Matrix, Beta-tricalcium phosphate
MeSH Terms: conditions — Periodontal Pocket

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mineralised Plasmatic Matrix Group (Experimental): Mineralized Plasmatic Matrix (MPM) is a product of mixing of two phases: the mineral phase and the plasma phase. After centrifugation, the white blood cells are recovered and mixed with the mineral phase of bone graft that can be autogenic, allogeneic bone, or a bone substitute like Xenogeneic Bone Synthetic. We will use Beta-tricalcium phosphate as a graft material. The result of this mixture is a homogeneous single component, which is compact and stable, containing the graft, the dense fibrin network, and the promoting healing. And then we are planning to place MPM material to extraction socket of impacted third molar tooth to improve periodontal healing at the distal aspect of second molar tooth. Additional after MPM places to extraction socket, Once the MPM has been placed, it will be covered with a Platelet Rich Fibrin (PRF) membrane and sutured as a primer.
  Interventions: Procedure: Impacted third molar surgery; Procedure: Application of mineralised plasmatic matrix
- Beta-tricalcium phosphate Group (Experimental): Beta-tricalcium phosphate graft will place in the extraction socket and cover with a PRF membrane.
  Interventions: Procedure: Impacted third molar surgery; Procedure: Application of β-tricalcium phosphate
- Control Group (Active Comparator): In the control group, after removal of impacted third molar tooth no material will be placed on the extraction socket. Only the extraction socket was primarily closed with non-resorbable sutures.
  Interventions: Procedure: Impacted third molar surgery

INTERVENTIONS:
Procedure: Impacted third molar surgery — Under local anesthesia, flap will be raised and mesioangular or horizontal impacted third molar tooth will be removed with routine technique. And then extraction socket will be irrigated with salin and will be primarily closed.
Procedure: Application of mineralised plasmatic matrix — After extraction of impacted third molar tooth, Mineralized Plasmatic Matrix will be placed to the socket as a graft material and will be covered with Platelet Rich Fibrin membrane. Then wound will be primarily closed.
  Other Names: Application platelet rich fibrin membrane
  Arms: Mineralised Plasmatic Matrix Group
Procedure: Application of β-tricalcium phosphate — After extraction of impacted third molar tooth, β-tricalcium phosphate will be placed to the socket as a graft material and will be covered with Platelet Rich Fibrin membrane. Then wound will be primarily closed.
  Other Names: Application platelet rich fibrin membrane
  Arms: Beta-tricalcium phosphate Group

SUMMARY:
This study evaluates the effectiveness of using Mineralized Plasmatic Matrix and β-tricalcium phosphate that placed to extraction socket as a graft material in terms of periodontal damage occurred in the distal aspect of the second molar after mandibular impacted third molar surgery.

ELIGIBILITY:
Inclusion Criteria:

* Medically healthy.
* Periodontally healthy patients.
* Patients with mesioangular or horizontal impacted teeth that will cause periodontal damage at the distal part of the second molar after surgery.

Exclusion Criteria:

* Crowns on second molar teeth.
* Poor oral hygiene.
* Patients with a systemic disease affecting periodontal healing.
* Pregnancy or lactation period.
* Patients undergoing orthodontic treatment.
* Smokers.
* The cases where the buccal or lingual cortical bone didn't remain intact following the extraction were also excluded.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-04-27 (Actual); Primary Completion 2020-05-20 (Estimated); Study Completion 2020-08-20 (Estimated)

PRIMARY OUTCOMES:
Periodontal pocket depth | At 0 day
  Initial periodontal pocket depth measurement at the distal aspect of second molar tooth before extraction.
Alveolar bone level | At 0 day
  Initial bone level measurement at the distal aspect of second molar tooth before extraction.

SECONDARY OUTCOMES:
Periodontal pocket depth | At 6th month
  Secondary measurement of periodontal pocket depth after extraction
Alveolar bone level | At 6th month
  Secondary measurement of bone level after extraction

CONTACTS AND LOCATIONS:
Overall Officials: Kubilay Işık, Study Chair — Consultant; Ali Kılınç, Study Director — Care Provider
Locations (1):
- Necmettin Erbakan University, Faculty of dentistry, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No